CLINICAL TRIAL: NCT02213744
Title: A Randomized, Multicenter, Open Label Study of MM-302 Plus Trastuzumab vs. Chemotherapy of Physician's Choice Plus Trastuzumab in Anthracycline Naive Patients With Locally Advanced/Metastatic HER2-Positive Breast Cancer
Brief Title: MM-302 Plus Trastuzumab vs. Chemotherapy of Physician's Choice Plus Trastuzumab in HER2-Positive Locally Advanced/Metastatic Breast Cancer Patients
Acronym: HERMIONE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Felt not to show benefit over control per DMC and confirmed via futility analysis
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-302-02-02-03
Record Dates: First submitted 2014-08-06; First posted 2014-08-11 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer; HER2 Positive Breast Cancer
Keywords: HER2-positive; HER2+; HER2; Locally Advanced Breast Cancer; Metastatic Breast Cancer; trastuzumab; Herceptin; pertuzumab; ado-trastuzumab emtansine; TDM-1; Perjeta; Kadcyla
MeSH Terms: conditions — Breast Neoplasms | interventions — gancotamab; Gemcitabine; Capecitabine; Vinorelbine; Trastuzumab

ARMS (2):
- MM-302 + trastuzumab (Experimental): MM-302 + trastuzumab
  Interventions: Drug: MM-302; Drug: Trastuzumab
- Chemotherapy of Physician's Choice plus trastuzumab (Active Comparator): Chemotherapy limited to one of the following: Gemcitabine, Capecitabine or Vinorelbine
  Interventions: Drug: Gemcitabine; Drug: Capecitabine; Drug: Vinorelbine; Drug: Trastuzumab

INTERVENTIONS:
Drug: MM-302
  Arms: MM-302 + trastuzumab
Drug: Gemcitabine
  Other Names: Gemzar
  Arms: Chemotherapy of Physician's Choice plus trastuzumab
Drug: Capecitabine
  Other Names: Xeloda
  Arms: Chemotherapy of Physician's Choice plus trastuzumab
Drug: Vinorelbine
  Arms: Chemotherapy of Physician's Choice plus trastuzumab
Drug: Trastuzumab
  Other Names: Herceptin

SUMMARY:
This study is an open label, randomized, multicenter trial of MM-302 plus trastuzumab. The trial is designed to demonstrate whether MM-302 plus trastuzumab is more effective than the chemotherapy of physician's choice (CPC) plus trastuzumab in locally advanced/metastatic HER2-positive breast cancer patients. Patients may not have been previously treated with an anthracycline in any setting. Patients must have received prior treatment with trastuzumab in any setting, have either progressed or are intolerant to ado-trastuzumab emtansine in the metastatic or locally advanced setting, have either progressed or are intolerant to pertuzumab in the metastatic or locally advanced setting or had disease recurrence within 12 months of pertuzumab treatment in the neoadjuvant or adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive cancer of the breast
* Patients must have documented locally advanced/metastatic disease, defined by the investigator, which is not amenable to resection with curative intent.
* Patients must have HER2-positive breast cancer as defined by ASCO/CAP 2013 guidelines that is confirmed by a Sponsor-designated central laboratory
* Patients must have progressed on, or be intolerant to pertuzumab in the LABC/MBC setting or had disease recurrence within 12 months of pertuzumab treatment in the neoadjuvant or adjuvant setting.
* Patients must have progressed on, or be intolerant to ado-trastuzumab emtansine in the LABC/MBC setting
* Patients must have been previously treated with trastuzumab in any setting (which may have been previously administered with or without pertuzumab)
* ECOG Performance Status of 0 or 1

Exclusion Criteria:

* Patients who have previously been treated with doxorubicin, liposomal doxorubicin, epirubicin, mitoxantrone, or any other anthracycline derivative
* Subjects with central nervous system (CNS) metastases, unless they have been treated and are stable without symptoms for 4 weeks after completion of treatment and must be off steroids for at least 4 weeks prior to enrollment
* Patients with any class of New York Heart Association (NYHA) CHF or heart failure with preserved ejection fraction (HFPEF)
* Patients with a history of known coronary artery disease or a myocardial infarction within the last 12 months
* Patients with a known history of serious cardiac arrhythmias requiring treatment (exception: controlled atrial fibrillation, paroxysmal supraventricular tachycardia)
* Patients who previously discontinued trastuzumab due to unacceptable cardiac toxicity
* Patients with a history of LVEF decline to below 50% during or after prior trastuzumab/lapatinib or other HER2 directed therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Independently assessed progression-free survival according to modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Approximately 2 years

SECONDARY OUTCOMES:
Locally assessed progression-free survival according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Approximately 2 years
Overall Survival | Approximately 3 years
Time to Treatment Failure | Approximately 2 years
Objective Response Rate based on independent and investigator review of tumor assessments | Approximately 2 years
Duration of Response (DoR) based on independent and investigator review of tumor assessments | Approximately 2 years
Safety | Approximately 2 years
  We will look specifically at the Number of Participants with Adverse Events related to MM-302 as compared to the control arm
Pharmacokinetic exposure of MM-302 | Approximately 2 years
  Area Under Curve (AUC) Time Frame: Cycles 1 and 2 - pre-infusion, post-infusion, and 168 hours post-dose. An optional timepoint at 8-96 hours post infusion is included during both cycles as well.

CONTACTS AND LOCATIONS:
Locations (109):
- United States (70):
  - Palo Verde Cancer Center, Glendale, Arizona
  - Mayo Clinic Cancer Center, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - St. Jude Heritage Healthcare, Fullerton, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Cancer Care Associates Medical Group, Redondo Beach, California
  - UCSF Medical Center, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Kaiser Permanent Medical Center, Vallejo, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Smilow Cancer Hospital at Yale New Haven Hospital, New Haven, Connecticut
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Florida Cancer Specialists & Research Institute, Fort Meyers, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Sarah Cannon Research Institute, New Port Richey, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - University of Miami Comprehensive Cancer Center, Plantation, Florida
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Northwestern University- Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - McFarland Clinic PC, Ames, Iowa
  - Johns Hopkins Medicine- The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, Coon Rapids, Minnesota
  - University of Minnesota- Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Morton Coleman MD, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Office of Carey K. Anders, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - St. Charles Health System, Bend, Oregon
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Bon Secours Saint Francis Hospital Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology- Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology- Medical City, Dallas, Texas
  - Texas Oncology, El Paso, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology-Houston Memorial City, Houston, Texas
  - The University of Texas- MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Oncology Associate, Norfolk, Virginia
  - Swedish Medical Center, Issaquah, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Austria (3):
  - Medizinische Universitat Innsbruck, Innsbruck
  - AKh Allgemeines Krankenhaus der Stadt Linz, Linz
  - Medical University of Vienna, Vienna
- Belgium (4):
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Antwerp
  - University Hospital Antwerp, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Clinique Saint-Joseph, Liège
- Canada (4):
  - London Regional Cancer Center, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University of Alberta- Cross Cancer Institute, Edmonton
  - McGill University Health Center, Québec
- Motol University Hospital, Prague, Czechia
- France (5):
  - Institut de Cancerologie de l'Ouest site Paul Papin, Angers
  - Centre Léon Bérard, Lyon
  - Hopital de l'Institut Curie, Paris
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
- Germany (3):
  - Universitatsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Interdisziplinares Onkologisches Zentrum, Munich
- Italy (9):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Centro Riferimento Oncologico, IRCCS, Istituto Nazionale Tumori, Aviano
  - Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremina
  - Oncology Unit Macerata Hospital, Macerata
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori, IRCCS Fondazione G. Pascale, Napoli
  - Instituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero S. Maria di Terni, Terni
- Spain (10):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Clinico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - H.U.Son Espases, Palma de Mallorca
  - Hospital de Navarra, Pamplona
  - Hospital Universitario Virgen de la Macarena, Seville

REFERENCES:
- [Derived] Miller K, Cortes J, Hurvitz SA, Krop IE, Tripathy D, Verma S, Riahi K, Reynolds JG, Wickham TJ, Molnar I, Yardley DA. HERMIONE: a randomized Phase 2 trial of MM-302 plus trastuzumab versus chemotherapy of physician's choice plus trastuzumab in patients with previously treated, anthracycline-naive, HER2-positive, locally advanced/metastatic breast cancer. BMC Cancer. 2016 Jun 3;16:352. doi: 10.1186/s12885-016-2385-z. PMID 27259714